CLINICAL TRIAL: NCT03946774
Title: Acute Effects of Dietary Protein on Monocyte/Macrophage mTOR Signaling and Downstream Sequela
Brief Title: Dietary Protein and Monocyte/Macrophage Mammalian Target of Rapamycin (mTOR) Signaling
Acronym: mTOR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Temporarily paused due to COVID-19 and expected to resume. This is not a suspension of IRB approval. PI has left the institution.
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 201808084
Record Dates: First submitted 2019-03-12; First posted 2019-05-13 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Dietary Protein
Keywords: Atherosclerosis; Macrophage/monocyte; mTOR; Autophagy; Apoptosis; Inflammation
MeSH Terms: conditions — Atherosclerosis; Inflammation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High protein (Active Comparator): Subjects getting high protein shake
  Interventions: Dietary Supplement: Dietary protein shake
- Low protein (Active Comparator): Subjects getting low protein shake
  Interventions: Dietary Supplement: Dietary protein shake

INTERVENTIONS:
Dietary Supplement: Dietary protein shake — It is a milk based protein shake. Ingredients include a combination of the following depending on protein content: Boost Plus (a commercial supplement), Unjury (a commercial whey protein isolate), nonfat dry milk powder, Sol Carb (commercial supplement composed of a carbohydrate polymer), canola oil, and water.
  In order to ensure consistency across all participants each beverage will be prepared in the Clinical Translational Research Unit Metabolic Kitchen under the supervision of a registered dietitian prior to the study participant's visit. Ingredients are individually weighed on a food scale by metabolic kitchen staff to the nearest 0.1 g and then mixed using a magnetic stir plate.
  Nutritional breakdown of the smoothies (high versus low protein):
  High protein drink nutrition: 500 kcal per serving, 50% protein, 17% fat, and 36% carbohydrate.
  Low (standard) protein drink nutrition: 500 kcal per serving, 10% protein, 17% fat, and 73% carbohydrate.

SUMMARY:
High protein low carbohydrate diets have become popular in recent years to help facilitate weight loss. It is controversial if these diets are associated with an increased risk of cardiovascular disease.

The investigators propose to administer high and low protein shakes to participants and measure effects on circulating monocytes, immune cells critical to the development of atherosclerosis and cardiovascular disease. In order to study circulating monocytes, blood will be collected from the study participants just prior to drinking the shake, and then 1 and 4 hours after drinking the shake.

In order to assess functional effects on monocytes, investigators will perform a series of assays comparing the results between individuals who drank high protein vs low protein shakes.

DETAILED DESCRIPTION:
Cardiovascular disease remains the leading cause of death globally with obesity as of one of the dominant modifiable risk factors. Obesity is also a precursor to several other cardiovascular risk factors including hypertension, hyperlipidemia, and diabetes. Almost all weight loss efforts utilize dietary modification with high protein/low carbohydrate diets serving as one of the most popular approaches. Despite the metabolic benefits of high dietary protein, recent studies have raised a concerning association with increased risk of atherosclerosis and cardiovascular disease. Although this remains controversial, there is some animal data showing evidence of dietary protein's proatherogenic role. These data are correlative and no mechanistic studies have been undertaken.

The downstream events after protein ingestion involve digestion of the protein into amino acids, increases in blood amino acids, and distribution to target tissues. Mouse models have definitively shown that circulating monocytes and macrophages of arterial blood vessels are particularly sensitive to this amino acid load with robust activation of the mTOR (mammalian target of rapamycin) signaling pathway. This in turn leads to inhibition of essential degradative processes of the macrophage such as autophagy and promotes release of pro-inflammatory cytokines. Thus, macrophage function in vascular beds becomes pathogenic leading to atherogenesis and cardiovascular disease

The translation of these mechanistic studies in animal models to human is the next obvious step in this research. However, no studies have elucidated the mechanisms of monocyte activation and function following administration of high dietary protein in humans. The investigators propose a pilot study to bridge an important gap in translational research which will elucidate the mechanisms by which dietary protein affects human monocyte function and the risk of atherosclerotic plaque formation. Specifically, the investigators will evaluate the acute activation of mTOR signaling and downstream sequelae in circulating monocytes following the administration of protein shakes. This study will address the hypothesis that humans exposed to high dietary protein will have significantly higher post-prandial monocyte mTOR activation with concomitant development of impaired degradative capacity and a proinflammatory state.

An understanding of these mechanisms has broad implications in the evaluation and future therapeutic interventions of cardiovascular disease.

In addition, this can provide a valuable clinical tool for health care providers in educating patients on dietary changes to ameliorate cardiovascular risk.

ELIGIBILITY:
Inclusion Criteria:

1. 18+ years of age
2. Able to drink milk based protein shake

Exclusion Criteria:

1. Current Pregnancy
2. Any food allergies
3. Personal Hx of Diabetes
4. Personal Hx of Heart Disease
5. Personal Hx of High blood pressure
6. Personal Hx of Stroke
7. Personal Hx of Cancer
8. Personal Hx of Organ transplant
9. Taking Rapamycin/Sirolimus
10. Taking Torisel/Temsirolimus
11. Taking Afinitor/Everolimus
12. Taking any statin medication (eg.simvastatin/atorvastatin/rosuvastatin etc)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-05-04 (Actual); Study Completion 2023-05-04 (Actual)

PRIMARY OUTCOMES:
Determination of amino acid levels and mTOR activation in circulating monocytes isolated from subjects ingesting high vs low protein drinks. | 0 Hour, 1 Hour, and 3 Hours
  Changes in amino acid levels and corresponding changes in mTOR activation will be quantified at baseline (time 0 hour prior to ingestion of a protein shake), then at 1 and 3 hours after ingestion of a protein shake.

SECONDARY OUTCOMES:
Determination of changes in autophagy and apoptosis markers in circulating monocytes over time after ingestion of a protein shake | 0 Hour, 1 Hour and 3 Hours
  Blood collected at three different time points (0, 1 and 3 hours) will be used to measure changes in markers of autophagy and apoptosis at baseline (time 0 hour prior to ingestion of a protein shake), then at 1 and 3 hours after ingestion of a protein shake.
Determination of changes in reactive oxygen species in circulating monocytes over time after ingestion of a protein shake. | 0 Hour, 1 Hour, and 3 Hours
  Blood collected at three different time points (0, 1 and 3 hours) will be used to measure changes in levels of reactive oxygen species at baseline (time 0 hour prior to ingestion of a protein shake), then at 1 and 3 hours after ingestion of a protein shake.
Determination of changes in inflammatory markers in circulating monocytes over time after ingestion of a protein shake. | 0 Hour, 1 Hour, and 3 Hours
  Blood collected at three different time points (0, 1 and 3 hours) will be used to measure changes in cytokines at baseline (time 0 hour prior to ingestion of a protein shake), then at 1 and 3 hours after ingestion of a protein shake.

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No